CLINICAL TRIAL: NCT03159117
Title: A Phase I Open-Label Dose Escalation of GD3 ADC (Pfizer PF-06688992) in Subjects With Unresectable Stage III or Stage IV Malignant Melanoma (B802WI209568)
Brief Title: Pfizer PF-06688992 in Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-165
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Melanoma
Keywords: GD3 ADC (Pfizer PF-06688992); Stage III Melanoma; Stage IV Melanoma; 17-165
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: This is a Phase 1 non-randomized, open-label, single-center, single-arm multiple dose escalation
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF 06688992 (Experimental): This clinical study will be a dose-finding phase I study in which patients will be treated with various doses of Pfizer PF-06688992 using a Bayesian dose escalation scheme.
  Interventions: Drug: PF-06688992

INTERVENTIONS:
Drug: PF-06688992 — (PF-06688992) will be administered on Day 1 of each 21-day cycle per the Dose Preparation and Administration Instructions (DAI) located in the Investigational Product Manual (Appendix 4Appendix 3) as an IV infusion over approximately 60 minutes. A cycle is defined as the time from Day 1 dose to the next Day 1 dose. If there are no treatment delays, a cycle will be 21 days. Each patient may receive PF-06688992 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination
  Other Names: GD3 ADC

SUMMARY:
The purpose of this research study is to learn about the safety and effectiveness of the study drug, PF-06688992. Before this study, PF-06688992 has never been given to people.

PF-06688992 is a targeted therapy for people with cancer. The investigators linked a chemotherapy drug to an antibody (protein found in the blood). The antibody will connect to GD3 which is found on most melanomas but on very few other cells in the body. The investigators hope that in this way, it will deliver this chemotherapy directly to the melanoma and not to normal tissues.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of melanoma confirmed at MSKCC
* Measurable unresectable Stage III or IV Malignant Melanoma and Response Criteria in Solid Tumors [RECIST], Version 1.1.
* Patients must have progressed on prior approved checkpoint inhibitor therapy, not tolerated approved checkpoint inhibitor therapy, or have a contraindication to approved checkpoint inhibitors. Patients with stable disease after approved checkpoint inhibitor therapy will also be eligible.
* Patients whose melanomas harbor a BRAF V600E or V600K mutation must have progressed on a RAF inhibitor. Patients who had to discontinue RAF inhibitor therapy because of toxicity but who did not progress will be eligible unless they responded to therapy. In that case, they will not be eligible unless they progress.
* Age ≥ 18 years
* ECOG performance status 0-1.
* Adequate Bone Marrow Function as defined by:

  °≥1,500/mm^3 or ≥ 1.5 x 10^9/L;
  * Platelets ≥ 100,000/mm3 or ≥ 100 x 109/L;
  * Hemoglobin ≥ 9 g/dL.
* Adequate Renal Function as defined by:

  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN); or
  * Estimated creatinine clearance ≥ 60 mL/min as calculated using the method standard for the institution.
* Adequate Liver Function as defined by:

  * Total serum bilirubin ≤ 1.5 x ULN unless the patient has documented Gilbert syndrome;
  * Aspartate and Alanine Aminotransferase (AST & ALT) ≤ 2.5 x ULN; ≤ 5.0 x ULN if there is liver involvement secondary to tumor;
  * Alkaline phosphatase ≤ 2.5 x ULN; (≤ 5 x ULN in case of bone metastasis).
* QTc interval < 470 msec.
* Recovery from all prior surgical or adjuvant treatment-related toxicities, to Baseline status, or a CTCAE Grade of 0 or 1, except for toxicities not considered a safety risk, such as alopecia. Post-surgical pain will not be considered a basis for exclusion.
* Negative serum/urine pregnancy test (for women of childbearing potential).
* Male and female patients of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 28 days after the last dose of assigned treatment. A patient is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.
* Evidence of a signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
* Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

* Patients with known symptomatic brain metastases requiring steroids.
* Patients with previously diagnosed brain metastases are eligible as long as they do not require CNS-directed therapy (including corticosteroids). If the patient has had radiation therapy or surgery, then they should have completed treatment and have discontinued corticosteroids for at least 2 weeks and must be neurologically stable.
* Patients with uveal melanoma will not be eligible as these tumors show low expression of GD3.
* Major surgery, radiation therapy or systemic anti-cancer therapy within 2 weeks of starting study treatment.
* Presence of ≥ Grade 2 peripheral neuropathy.
* Significant prior infusion reaction to monoclonal antibodies that required treatment with systemic steroids.
* Active and clinically significant bacterial, fungal or viral infection.

  * Known infections with hepatitis B (HBV) or hepatitis C (HCV),
  * Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness not controlled (with undetectable viral load) on HAART therapy. Patients on HAART with undetectable viral loads may be eligible per PI judgment.
* Pregnant or breastfeeding; males and females of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after last dose of investigational product.
* Patients currently receiving active treatment for melanoma.
* Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack.
* Any ongoing cardiac dysrhythmias of NCI CTCAE Grade >2, NCI CTCAE Grade 4 atrial fibrillation, or QTcF interval >470 msec, except for documented Right Bundle Branch Block, at screening.
* Chronic Bronchitis or Emphysema requiring oxygen therapy within the last 6 months.
* Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality or uncontrolled hypertension that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
the Recommended Phase 2 Dose | 1 year
  using a Bayesian dose escalation scheme

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm